CLINICAL TRIAL: NCT02683889
Title: The Use of Acthar (ACTH) in Patients With Focal Segmental Glomerulosclerosis (FSGS) Who Have Developed Chronic Kidney Disease Stage V (CKD) or End Stage Renal Disease (ESRD) and Are Undergoing a Renal Transplant
Brief Title: Use of Acthar in Patients With FSGS That Will be Undergoing Renal Transplantation
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-2336
Record Dates: First submitted 2016-02-05; First posted 2016-02-17 (Estimated); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: FSGS
Keywords: Kidney transplant
MeSH Terms: interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- One arm (Experimental): One arm will receive acthar to measure rate of recurrence of FSGS after transplant. There are no other arms. We do have previous data that FSGS recurs in 23% of kidney transplants.
  Interventions: Drug: Acthar

INTERVENTIONS:
Drug: Acthar — patients will receive acthar 80 units twice a week for 6 months and will measure recurrence of FSGS

SUMMARY:
This study will evaluate the use of Acthar in patients to undergo renal transplantation and will measure the rate of FSGS recurrence.

DETAILED DESCRIPTION:
This is a prospective study enrolling renal transplant recipients with the primary native kidney disease of FSGS.

Primary endpoint is rate of recurrence of FSGS as seen in renal transplant biopsies and in rate of proteinuria. Secondary endpoint is renal function after transplantation The target subject number is 20 patients and the target population is primary FSGS patients. By the current data, FSGS should recur in 23% of patients. Therefore, it would be expected that at least 4 patients will develop recurrent FSGS after renal transplantation.

Screening will be performed by the Principal Investigator during the kidney transplant evaluation clinics and during the wait list kidney transplant evaluation clinic. All patients with FSGS will have maintenance immunosuppression with belatacept (if EBV positive), prograf, cellcept and prednisone. If after one year the patient has been stable and there has not been rejection, will stop the prograf and continue solely with belatacept, cellcept and prednisone.

Dosage and Administration of Acthar The dose of acthar to be given to every enrolled patient will be 80 units twice a week for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* FSGS
* To receive either a live donor or deceased donor kidney transplant

Exclusion Criteria:

* Not having FSGS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrence of FSGS as seen in renal transplant biopsies proteinuria | 2 years
  This will be studied in the renal transplant biopsies
Rate of recurrence of proteinuria | 2 years
  By measurement of urine protein and urine creatinine ratio

SECONDARY OUTCOMES:
renal function after transplantation | 1 year
  By measurement of the estimated glomerular filtration rate with patient's creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Sixto Giusti, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Medstar Georgetown Transplant Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT02683889/Prot_SAP_000.pdf